CLINICAL TRIAL: NCT04329559
Title: Clinical Characteristics of COVID-19 in Patients With Pre-existing Cirrhosis (COVID-Cirrhosis-CHESS2002): A Multicentre Observational Study
Brief Title: COVID-19 in Patients With Pre-existing Cirrhosis (COVID-Cirrhosis-CHESS2002): A Multicentre Observational Study
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); LanZhou University (Other); Minda Hospital Affiliated to Hubei University for Nationalities (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture (Other); Tianjin Second People's Hospital (Other); The Sixth People's Hospital of Shenyang (Other); Guangxi Zhuang Autonomous Region (Unknown); Shenzhen Third People's Hospital (Other); Ankang Central Hospital (Other); Xingtai People's Hospital (Other); Dalian Sixth People's Hospital (Unknown); The Central Hospital of Lishui City (Other); The Affiliated Third Hospital of Jiangsu University (Unknown); Suizhou Hospital, Hubei University of Medicine (Unknown)
Responsible Party: Principal Investigator, Xiaolong Qi, Chief, Institute of Portal Hypertension, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2002
Record Dates: First submitted 2020-03-29; First posted 2020-04-01 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: COVID-19; Liver Cirrhosis
Keywords: COVID-19; Liver cirrhosis; Clinical outcome
MeSH Terms: conditions — COVID-19; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 pandemic with SARS-CoV-2 infection has become a global challenge. Though most cases of COVID-19 are mild, the disease can also be fatal. Patients with liver cirrhosis are more susceptible to damage from SARS-CoV-2 infection considering their immunocompromised status. The spectrum of disease and factors that influence the disease course in COVID-19 cases with liver cirrhosis are incompletely defined. This muilticentre observational study (COVID-Cirrhosis-CHESS2002) aims to study the clinical characteristics and risk factors associated with specific outcomes in COVID-19 patients with pre-existing liver cirrhosis.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) pandemic with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection has become a global challenge. Though most cases of COVID-19 are mild, the disease can also be fatal. Patients with liver cirrhosis are more susceptible to damage from SARS-CoV-2 infection considering their immunocompromised status. The spectrum of disease and factors that influence the disease course in COVID-19 cases with liver cirrhosis are incompletely defined. This muilticentre observational study (COVID-Cirrhosis-CHESS2002) aims to study the clinical characteristics and risk factors associated with specific outcomes in COVID-19 patients with pre-existing liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged 18 or above;
* 2) Laboratory-confirmed COVID-19 infection;
* 3) Pre-existing liver cirrhosis based on liver biopsy or clinical findings.

Exclusion Criteria:

* 1) Pregnancy or unknown pregnancy status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19 infection with pre-existing liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
All-cause mortality of COVID-19 patients with liver cirrhosis | From illness onset of COVID-19 to death from any cause, up to 365 days
  7-day, 28-day, 60-day, 180-day and 365-day all-cause mortality of COVID-19 patients with liver cirrhosis

SECONDARY OUTCOMES:
Liver-related mortality of COVID-19 patients with liver cirrhosis | From illness onset of COVID-19 to death from liver-related cause, up to 365 days
  7-day, 28-day, 60-day, 180-day and 365-day liver-related mortality of COVID-19 patients with liver cirrhosis
Risk factors associated with specific outcomes of COVID-19 patients with liver cirrhosis | From hospital admission to death, up to 365 days
  Risk factors (laboratory findings, imaging findings, etc.) associated with specific outcomes (death, etc.) of COVID-19 patients with liver cirrhosis
Baseline characteristics of COVID-19 patients with liver cirrhosis | 1 Day
  Baseline characteristics (laboratory findings, imaging findings, etc.) of COVID-19 patients with liver cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Chen, MD, Study Chair — Renmin Hospital of Wuhan University; Xiaolong Qi, MD, Study Chair — LanZhou University; Fengmei Wang, MD, Principal Investigator — Tianjin Second People's Hospital; Ye Gu, MD, Principal Investigator — The Sixth People's Hospital of Shenyang; Zicheng Jiang, MD, Principal Investigator — Ankang Central Hospital; Guo Zhang, MD, Principal Investigator — Guangxi Zhuang Autonomous Region; Yong Zhang, MD, Principal Investigator — Dalian Sixth People's Hospital; Dengxiang Liu, MD, Principal Investigator — Xingtai People's Hospital; Qing He, MD, Principal Investigator — Shenzhen Third People's Hospital; Hua Yang, MD, Principal Investigator — Minda Hospital Affiliated to Hubei University for Nationalities; Zhengyan Wang, MD, Principal Investigator — Suizhou Hospital, Hubei University of Medicine; Bin Xiong, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Xiaodan Li, MD, Principal Investigator — The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture; Hongguang Zhang, MD, Principal Investigator — The Affiliated Third Hospital of Jiangsu University; Chuxiao Shao, MD, Principal Investigator — The Central Hospital of Lishui City; Hongmei Yue, MD, Principal Investigator — LanZhou University
Locations (15):
- China (15):
  - Dalian Sixth People's Hospital, Dalian
  - Minda Hospital Affiliated to Hubei University for Nationalities, Enshi
  - The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture, Enshi
  - The First Hospital of Lanzhou University, Lanzhou
  - The Central Hospital of Lishui City, Lishui
  - Guangxi Zhuang Autonomous Region, Nanning
  - The Sixth Peoples Hospital of Shenyang, Shenyang
  - Shenzhen Third People's Hospital, Shenzhen
  - Suizhou Hospital, Hubei University of Medicine, Suizhou
  - Tianjin Second People's Hospital, Tianjin
  - Ankang Central Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuhan Union Hospital, Wuhan
  - Xingtai People's Hospital, Xingtai
  - The Affiliated Third Hospital of Jiangsu University, Zhenjiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Zhang C, Shi L, Wang FS. Liver injury in COVID-19: management and challenges. Lancet Gastroenterol Hepatol. 2020 May;5(5):428-430. doi: 10.1016/S2468-1253(20)30057-1. Epub 2020 Mar 4. No abstract available. PMID 32145190
- [Background] Bangash MN, Patel J, Parekh D. COVID-19 and the liver: little cause for concern. Lancet Gastroenterol Hepatol. 2020 Jun;5(6):529-530. doi: 10.1016/S2468-1253(20)30084-4. Epub 2020 Mar 20. No abstract available. PMID 32203680
- [Background] Xu L, Liu J, Lu M, Yang D, Zheng X. Liver injury during highly pathogenic human coronavirus infections. Liver Int. 2020 May;40(5):998-1004. doi: 10.1111/liv.14435. Epub 2020 Mar 30. PMID 32170806